CLINICAL TRIAL: NCT03971123
Title: A Phase 1, Randomised, Single-center, Single-dose, Placebo-controlled, 3-Way Crossover Study to Compare the Pharmacokinetics, Safety and Tolerability of a Lipid Multi-particulate (LMP) Formulation and Spray-dried (SD) Formulations of Tricaprilin (TC) on Ketone Body Production (Part 1). Addendum to Include a 2-way Crossover to Compare the Pharmacokinetics, Safety and Tolerability of Two Spray-dried (SD) Formulations of Tricaprilin (TC) on Ketone Body Production (Part 2)
Brief Title: Study to Compare the Pharmacokinetics of Tricaprilin Formulations and a Placebo on Ketone Body Production
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cerecin (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: AC-19-017
Record Dates: First submitted 2019-05-27; First posted 2019-06-03 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — tricaprylin; AC-1202

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- AC-SD-03 (for Part 1) (Experimental): Tricaprilin SD formulation, single dose (20g tricaprilin). Administered orally.
  Interventions: Drug: Tricaprilin
- AC-LMP-01 (for Part 1) (Experimental): Tricaprilin LMP formulation, single dose (20g tricaprilin). Administered orally.
  Interventions: Drug: Tricaprilin
- AC-SD-03P (for Part 1) (Experimental): Placebo formulation, single dose. Administered orally
  Interventions: Drug: Placebo
- AC-1202 (for Part 2) (Experimental): Tricaprilin SD formulation, single dose (20g caprylic triglyceride). Administered orally.
  Interventions: Drug: Tricaprilin
- AC-SD-03 (for Part 2) (Experimental): Tricaprilin SD formulation, single dose (20g tricaprilin). Administered orally.
  Interventions: Drug: Tricaprilin

INTERVENTIONS:
Drug: Tricaprilin — Tricaprilin formulated as AC-SD-03 50g of AC-SD-03 (20g tricaprilin) mixed in 240mL dosing liquid at Hour 0 Day 1
  Other Names: AC-SD-03
  Arms: AC-SD-03 (for Part 1); AC-SD-03 (for Part 2)
Drug: Tricaprilin — Tricaprilin formulated as AC-LMP-01 50g of AC-LMP-01 (20g tricaprilin) mixed in 240mL dosing liquid at Hour 0 Day 1
  Other Names: AC-LMP-01
  Arms: AC-LMP-01 (for Part 1)
Drug: Placebo — Matching placebo to AC-SD-03 50g of AC-SD-03P mixed in 240mL dosing liquid at Hour 0 Day 1
  Other Names: AC-SD-03P
  Arms: AC-SD-03P (for Part 1)
Drug: Tricaprilin — Tricaprilin formulated as AC-1202 60g of AC-1202 (20g caprlic triglyceride) mixed in 240mL dosing liquid at Hour 0 Day 1
  Other Names: AC-1202
  Arms: AC-1202 (for Part 2)

SUMMARY:
Phase 1, Single-center, Open-label Study, Healthy Adult Male Subjects.

Part 1:Single-dose, Placebo-controlled, 3-Way Crossover PK Study

Part 2: Single dose 2-way comparator PK Study

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male 18 - 50 years of age, inclusive, at Screening.
* Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m2 at Screening.
* Agrees to comply with study procedures.
* Continuous non smoker who has not used nicotine containing products or smoking no more than 10 cigarettes per week for at least 3 months prior to Screening and will not use them throughout the study.
* A non-vasectomized subject must agree to use a condom or abstain from sexual intercourse during the study. No restrictions are required for a vasectomized male provided his vasectomy has been performed 4 months or more prior to Screening. A subject who has been vasectomized less than 4 months prior to Screening must follow the same restrictions as a non-vasectomized male.
* Subject is able and willing to consume a prescribed full breakfast on at least 3 occasions. Subject does not have specific dietary requirements (vegetarian, vegan, lactose-free, low-fat, etc.).
* Subject is not consuming a ketogenic diet (defined by consumption of < 50 gm carbohydrates per day).
* Has given voluntary, written informed consent to participate in the study.
* For Cohort 1, the Chinese subjects are restricted to being of Chinese heritage (irrespective of country of residence) and defined as all 4 grandparents of the subject must be Chinese (for Part 1 only).

Exclusion Criteria:

* History or presence of alcoholism or substance abuse disorder within the last year.
* Positive urine drug screen at Screening or Check-in.
* Subject is currently actively using MCTs, ketone esters, or other ketogenic products or is following a ketogenic diet.
* Clinically significant abnormal laboratory results at Screening.
* Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to dosing, administration of a biological product in the context of a clinical research study within 90 days prior to dosing, or concomitant participation in an investigational study involving no drug or device administration.
* Subject has a known allergy to the study drug's active or inactive ingredients.
* Subject has been following a ketogenic diet (or other diet incompatible with the on-study diet), in the opinion of the investigator.
* Unable to refrain from, or anticipates the use of, any drug including prescription and non-prescription medications, herbal remedies or vitamin supplements beginning 14 days prior to the first dose and throughout the study, unless deemed acceptable by the PI. Paracetamol (up to 4g per 24-hour period) or ibuprofen (up to 1,200 mg per 24-hour period) may be permitted during the study.
* Has had alcohol 48 hours prior to Day -1 of Period 1.
* Any other condition which, in the investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-08-30 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2020-05-26 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single-dose administration of each of tricaprilin formulations and the placebo formulation, in healthy, male volunteers (for Part 1 and 2) | 11 days
  Number of subjects with treatment related adverse events as assessed by CTCAE
Pharmacokinetics (PK) parameters of Total Ketones, Tricaprilin and Octanoic acid levels after single dose of each of tricaprilin formulations and the placebo formulation using AUC(0-t) (for Part 1 and 2) | 1 day
  AUC(0-t) will be calculated from PK concentrations of Total Ketones (B-hydroxybutyrate and Acetoacetate), Tricaprilin and Octanoic Acid Levels. AUC (0-t) = Area under the concentration-time curve from 0 to last quantifiable concentration. Summary statistics will be generated for each PK parameter.
Pharmacokinetics (PK) parameters of Total Ketones, Tricaprilin and Octanoic acid levels after single dose of each of tricaprilin formulations and the placebo formulation using Cmax (for Part 1 and 2) | 1 day
  Cmax will be calculated from PK concentrations of Total Ketones (B-hydroxybutyrate and Acetoacetate), Tricaprilin and Octanoic Acid Levels. Cmax = Cmax is maximum concentration, determined directly from individual concentration-time data.Summary statistics will be generated for each PK parameter.
Pharmacokinetics (PK) parameters of Total Ketones, Tricaprilin and Octanoic acid levels after single dose of each of tricaprilin formulations and the placebo formulation using Tmax (for Part 1 and 2) | 1 day
  Tmax will be calculated from PK concentrations of Total Ketones (B-hydroxybutyrate and Acetoacetate), Tricaprilin and Octanoic Acid Levels. Tmax = Time to reach maximum observed concentration, determined directly from individual concentration-time data.Summary statistics will be generated for each PK parameter.

SECONDARY OUTCOMES:
ApoE4 Genotyping (for Part 1 only) | 1 day
  The Apo-E test provides a value represented by the type of the allele (E2, E3,E4).The allelic variant of the Apo-E (APOE4) will be evaluated for effects on tricaprilin induced ketone body production.

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No